CLINICAL TRIAL: NCT01118026
Title: Phase II Trial of Response-Adapted Therapy Based on Positron Emission Tomography (PET) for Bulky Stage I and Stage II Classical Hodgkin Lymphoma (HL)
Brief Title: Response-Based Therapy Assessed By PET Scan in Treating Patients With Bulky Stage I and Stage II Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50801; CDR0000669076 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-02034 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; adult favorable prognosis Hodgkin lymphoma; adult lymphocyte depletion Hodgkin lymphoma; adult lymphocyte predominant Hodgkin lymphoma; adult mixed cellularity Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma; adult unfavorable prognosis Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — BEACOPP protocol; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABVD +/- BEACOPP + radiation (Experimental): Patients receive ABVD administered by intravenous (IV) infusion on days 1 and 15 of each cycle. A cycle is considered 28 days. Patients receive a total of two cycles.
  Patients undergo a PET scan following two cycles of ABVD. If the PET scan is negative, then the patient will receive four more cycles of ABVD (a total of 6 cycles of ABVD). If the PET scan is positive, then the patient receives four cycles of escalated BEACOPP for 21 days (a total of 4 cycles).
  3-6 weeks after BEACOPP therapy, patients receive radiation therapy for 5 days per week (a total of 3.5 weeks).
  All patients will be followed for a maximum of ten years.
  Interventions: Drug: ABVD; Drug: BEACOPP; Radiation: radiation therapy

INTERVENTIONS:
Drug: ABVD — doxorubicin 25 mg/m^2 IV bleomycin 10 units/m^2 IV vinblastine 6 mg/m^2 IV dacarbazine 375 mg/m^2 IV
Drug: BEACOPP — bleomycin 10 units/m^2 IV on Day 8 etoposide 200 mg/m^2 IV on Days 1, 2 and 3 doxorubicin 35 mg/m^2 IV on Day 1 cyclophosphamide 1250 mg/m^2 IV on Day 1 vincristine 1.4 mg/m^2 IV on Day 8 procarbazine 100 mg/m^2 orally on Days 1-7 prednisone 40 mg/m^2 orally on Days 1-14
Radiation: radiation therapy

SUMMARY:
This research is being done in order to improve treatment outcomes in patients diagnosed with bulky, early stage Hodgkin lymphoma and to reduce the side effects that are associated with use of radiation used in current treatments. The chemotherapy treatment in this study consists of a combination of four drugs approved by the Food and Drug Administration (FDA): doxorubicin, bleomycin, vinblastine, and dacarbazine. This regimen (called ABVD) has been found to be effective in treating patients with Hodgkin lymphoma and is considered the standard of treatment used with radiation therapy in patients with bulky early stage Hodgkin lymphoma. As part of the evaluation of the effectiveness of the chemotherapy treatment, PET scans will be obtained during the course of therapy. The usefulness of this PET scan will be evaluated to determine whether radiation may be left out in the treatment of disease if the PET scan shows that the patient has responded to chemotherapy alone. The plan is to identify a group of patients using early PET scans in order to change to a chemotherapy treatment called BEACOPP (bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine and prednisone). It is one of the most highly effective chemotherapy regimens for Hodgkin lymphoma, but is associated with more side effects than ABVD. Although it has become standard of care in Europe, its use has been more limited in the U.S. because of concerns about toxicity.

DETAILED DESCRIPTION:
This is single-arm phase II clinical trial of response-adapted therapy based on PET for bulky stage I and stage II Hodgkin lymphoma. A maximum of 123 patients will be entered to the study. The primary outcome of this study is progression-free survival (PFS), defined as the time from study entry to disease progression or death.

Primary Objective:

To determine the progression-free survival (PFS) at 36 months from enrollment for patients with bulky stage I and II Hodgkin lymphoma. All patients will begin treatment with ABVD. Patients who are PET negative after 2 cycles of chemotherapy will receive 6 cycles of ABVD without radiotherapy. Patients who are PET positive after 2 cycles of ABVD will then receive 4 cycles of escalated BEACOPP followed by IFRT. A comparison will be made of the 36-month PFS between patients who are PET positive and those who are PET negative following 2 cycles of ABVD.

Secondary Objectives:

1. To evaluate the complete response (CR) rate of patients diagnosed with bulky stage I and II Hodgkin lymphoma following PET response-adapted chemotherapy with or without radiation therapy.
2. To determine the predictive value of FDG uptake using various semiquantitative approaches, at baseline, after 2 cycles of ABVD and at completion of therapy.
3. To determine the predictive value of volumetric vs. 2 dimensional (2-D) measurement changes on CT between baseline and after 2 cycles, at the end of chemotherapy (PET negative patients only) and after RT (PET positive patients only) and compare with PET parameters.
4. To determine if changes in both qualitative and semiquantitative FDG-PET findings between baseline and after cycle 2, at end of chemotherapy (PET negative patients only) and after RT (PET positive patients only) with combination analyses with incorporating changes obtained from dedicated CT scans, correlate with response and PFS.
5. To compare the predictive value of both qualitative and semiquantitative FDG-PET changes, 2-D and volumetric CT changes, and combinatorial analyses (PET+dedicated CT data) with molecular parameters, and conventional parameters, including IPS.
6. To assess whether elevated baseline serum soluble CD30 (sCD30), IL10, CCL17, and CCL22 correlate with clinical response and PFS.
7. To assess whether persistent or recurrent elevation of serial serum sCD30, IL10, CCL17, or CCL22 correlate with relapse/progression or PET scan results.
8. To confirm independently useful tissue biomarkers (bcl-2, MAL, FOXP3, CD68, GzB) for risk stratification in patients with bulky stage I and II Hodgkin lymphoma treated with this regimen.
9. To compare mediastinal bulk on standing PA and lateral chest x-ray (> 0.33 maximum chest diameter) with chest CT (mass > 10 cm).

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 2-3 years, and then once a year for a maximum of ten years from the time of entry on the study.

ELIGIBILITY:
1. Documentation of Disease:

   * Histologically documented Hodgkin lymphoma subclassified according to the WHO modification of the Rye Classification and staged according to the modified Ann Arbor Staging Classification system.

     * Patients must have clinical stage IA, IB, IIA or IIB.
     * Patients with "E" extensions will be eligible if all other criteria have been met.
     * Nodular lymphocyte predominant Hodgkin lymphoma is excluded.
     * Core needle biopsies are acceptable if they contain adequate tissue for primary diagnosis and immunophenotyping. Fine needle aspirates are not acceptable. If multiple specimens are available, please submit the most recent. Failure to submit pathology materials within 60 days of patient registration will be considered a major protocol violation.
   * Patients must have a mediastinal mass > 0.33 maximum intrathoracic diameter on standing postero-anterior chest x-ray or mass measuring > 10 cm in its largest diameter.
2. Second Malignancy: No "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse.
3. Prior Therapy - Patients may have had one cycle only of ABVD prior to enrolling on study. No other prior treatment (chemotherapy or radiation therapy) for Hodgkin lymphoma is allowed. If patient has had one cycle of ABVD, in order to be eligible to enroll on CALGB 50801, the patient must have had all of the following tests prior to starting the first cycle of ABVD:

   * LVEF by ECHO or MUGA
   * PFTs (including DLCO/FVC)CT scan (neck*, chest, abdomen, pelvis)
   * FDG-PET/CT scan
   * Chest X-ray, PA & Lateral
   * CBC, differential, platelets
   * ESR
   * Serum creatinine
   * Glucose
   * AST
   * Alkaline phosphatase
   * Bilirubin
   * LDH

   Patients with a negative FDG-PET/CT scan do not need to have had a dedicated neck CT scan prior to starting the previous cycle of ABVD.
4. ECOG Performance status 0-2.
5. LVEF and DLCO - LVEF by ECHO or MUGA within institutional normal limits unless thought to be disease related. DLCO ≥ 60% with no symptomatic pulmonary disease unless thought to be disease related.
6. HIV Infection - Patients with known HIV must have a CD4 count > 350 and be on concurrent antiretrovirals. Patients with a history of intravenous drug abuse or any behavior associated with an increased risk of HIV infection should be tested for exposure to the HIV virus. An HIV test is not required for entry on this protocol, but is required if the patient is perceived to be at risk.
7. Pregnancy Restrictions - Non-pregnant and non-nursing. Due to the teratogenic potential of the agents used in this study, pregnant or nursing women may not be enrolled. Women and men of reproductive potential should agree to use an effective means of birth control.
8. Age Restricitions - Age 18 - 60 years
9. Initial Required Laboratory Data:

   * ANC ≥ 1000/μL
   * Platelet count ≥ 100,000/μL
   * Serum Creatinine ≤ 2 mg/dL
   * Bilirubin* ≤ 2 x upper limit of normal
   * AST ≤ 2 x upper limit of normal* - In the absence of Gilbert's disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann S. LaCasce, MD, Study Chair — Dana-Farber Cancer Institute
Locations (55):
- United States (55):
  - Naval Medical Center -San Diego, San Diego, California
  - Saint Helena Hospital, St. Helena, California
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Nashua, Nashua, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Weill Medical College of Cornell University, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Carolinas HealthCare System NorthEast, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] LaCasce AS, Dockter T, Ruppert AS, Kostakoglu L, Schoder H, Hsi E, Bogart J, Cheson B, Wagner-Johnston N, Abramson J, Blum K, Leonard JP, Bartlett NL. Positron Emission Tomography-Adapted Therapy in Bulky Stage I/II Classic Hodgkin Lymphoma: CALGB 50801 (Alliance). J Clin Oncol. 2023 Feb 10;41(5):1023-1034. doi: 10.1200/JCO.22.00947. Epub 2022 Oct 21. PMID 36269899
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/about-cancer/treatment/clinical-trials/search/v?id=NCI-2011-02034&q=CALGB-50801

RESULTS

PARTICIPANT FLOW:
Groups:
- ABVD +/- BEACOPP + Radiation: Patients receive ABVD administered by intravenous (IV) infusion on days 1 and 15 of each cycle. A cycle is considered 28 days. Patients receive a total of two cycles. > > Patients undergo a PET scan following two cycles of ABVD. If the PET scan is negative, then the patient will receive four more cycles of ABVD (a total of 6 cycles of ABVD). If the PET scan is positive, then the patient receives four cycles of escalated BEACOPP for 21 days (a total of 4 cycles). >
  > 3-6 weeks after BEACOPP therapy, patients receive radiation therapy for 5 days per week (a total of 3.5 weeks).>
  > All patients will be followed for a maximum of ten years.>
  > ABVD: doxorubicin 25 mg/m^2 IV> bleomycin 10 units/m^2 IV> vinblastine 6 mg/m^2 IV> dacarbazine 375 mg/m^2 IV>
  > BEACOPP: bleomycin 10 units/m^2 IV on Day 8> etoposide 200 mg/m^2 IV on Days 1, 2 and 3> doxorubicin 35 mg/m^2 IV on Day 1> cyclophosphamide 1250 mg/m^2 IV on Day 1> vincristine 1.4 mg/m^2 IV on Day 8> procarbazine 100 mg/m^2 orally on Days 1-7> prednisone 40 mg/m^2 orally on Days 1-14>
  > radiation therapy
Period: Overall Study
Arm/Group | ABVD +/- BEACOPP + Radiation
Started | 101
Completed | 101
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ABVD +/- BEACOPP + Radiation
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 87
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 36 Months
Description: Progression-free survival (PFS) is defined as the time from first PET/CT scan to disease progression or death. Patients who are alive without disease progression will be censored at the time of their most recent disease evaluation. The Kaplan-Meier three-year (36 month) survival estimates and confidence intervals are presented below.
Time Frame: Up to 36 months
Population: Six patients were not eligible for this analysis and one patient was not evaluated for PET status screening. All patients that were eligible and evaluated for PET screening were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ABVD (PET-negative): Patients receive ABVD administered by intravenous (IV) infusion on days 1 and 15 of each cycle. A cycle is considered 28 days. Patients receive a total of two cycles. > > Patients undergo a PET scan following two cycles of ABVD. If the PET scan is negative, then the patient will receive four more cycles of ABVD (a total of 6 cycles of ABVD). >
  >
  > All patients will be followed for a maximum of ten years.>
  > ABVD: doxorubicin 25 mg/m^2 IV> bleomycin 10 units/m^2 IV> vinblastine 6 mg/m^2 IV> dacarbazine 375 mg/m^2 IV
- ABVD + BEACOPP + Radiation (PET-positive): Patients receive ABVD administered by intravenous (IV) infusion on days 1 and 15 of each cycle. A cycle is considered 28 days. Patients receive a total of two cycles. > > Patients undergo a PET scan following two cycles of ABVD. If the PET scan is positive, then the patient receives four cycles of escalated BEACOPP for 21 days (a total of 4 cycles). >
  > 3-6 weeks after BEACOPP therapy, patients receive radiation therapy for 5 days per week (a total of 3.5 weeks).>
  > All patients will be followed for a maximum of ten years.>
  > ABVD: doxorubicin 25 mg/m^2 IV> bleomycin 10 units/m^2 IV> vinblastine 6 mg/m^2 IV> dacarbazine 375 mg/m^2 IV>
  > BEACOPP: bleomycin 10 units/m^2 IV on Day 8> etoposide 200 mg/m^2 IV on Days 1, 2 and 3> doxorubicin 35 mg/m^2 IV on Day 1> cyclophosphamide 1250 mg/m^2 IV on Day 1> vincristine 1.4 mg/m^2 IV on Day 8> procarbazine 100 mg/m^2 orally on Days 1-7> prednisone 40 mg/m^2 orally on Days 1-14>
  > radiation therapy
Arm/Group | ABVD (PET-negative) | ABVD + BEACOPP + Radiation (PET-positive)
Number analyzed (Participants) | 73 | 21
percentage of participants | 93.1 [87.4 to 99.1] | 89.7 [77.2 to 100]
Statistical Analysis 1: Comparison: ABVD (PET-negative) vs ABVD + BEACOPP + Radiation (PET-positive); Test type: Superiority; p = 0.9669, Log Rank

2. Secondary Outcome: Complete Response
Description: A Complete Response (CR) is defined as the complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. For this endpoint, the best response at any time post-baseline was analyzed
Time Frame: Up to 8 weeks
Population: All eligible patients patients who were screened for PET status and were evaluated for response are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ABVD (PET-negative) | ABVD + BEACOPP + Radiation (PET-positive)
Number analyzed (Participants) | 73 | 21
Participants | 73 | 16

3. Other Pre Specified Outcome: Comparison of Qualitative and Semiquantitative Fludeoxyglucose-PET Findings/Changes, 2-D and Volumetric CT Changes, and Combinatorial Analyses (PET + Dedicated CT Data) With Molecular Parameters and Conventional Parameters
Time Frame: Up to 3 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Volumetric vs 2-dimensional (2-D) Measurement Changes for Target Lesions Between Baseline and After Course 2, at the End of Chemotherapy, and After IFRT
Time Frame: Up to 3 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Determination of the Optimal Cutoff for Absolute Decrease in Maximum SUV Body Weight (SUVbw) and SUV Lean Body Mass (SUVlbm), Relative Uptake in Tumor vs Various Reference Anatomic Sites, IHP Criteria as Well as Various Cutoffs for Post-therapy Maxim ...
Time Frame: Up to 3 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Standard Uptake Values (SUVs) for Target Sites Measured at Baseline, After Course 2, and After Completion of Therapy
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 36 months
Groups:
- ABVD +/- BEACOPP + Radiation: radiation therapy
Arm/Group | ABVD +/- BEACOPP + Radiation
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 100/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABVD +/- BEACOPP + Radiation (N=100)
Anemia (Blood and lymphatic system disorders) | 75 (300)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (11)
Chest pain - cardiac (Cardiac disorders) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 7 (12)
Supraventricular tachycardia (Cardiac disorders) | 2 (4)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Cushingoid (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (4)
Dry eye (Eye disorders) | 2 (3)
Flashing lights (Eye disorders) | 1 (3)
Watering eyes (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 17 (19)
Bloating (Gastrointestinal disorders) | 6 (12)
Cheilitis (Gastrointestinal disorders) | 1 (4)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 49 (117)
Diarrhea (Gastrointestinal disorders) | 27 (45)
Dry mouth (Gastrointestinal disorders) | 6 (16)
Dyspepsia (Gastrointestinal disorders) | 17 (31)
Dysphagia (Gastrointestinal disorders) | 10 (12)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 3 (5)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 (12)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 4 (4)
Gingival pain (Gastrointestinal disorders) | 1 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 4 (8)
Mucositis oral (Gastrointestinal disorders) | 36 (61)
Nausea (Gastrointestinal disorders) | 83 (275)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (2)
Oral pain (Gastrointestinal disorders) | 13 (15)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 3 (7)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 5 (10)
Toothache (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 33 (61)
Chills (General disorders) | 9 (12)
Edema face (General disorders) | 2 (2)
Edema limbs (General disorders) | 9 (19)
Edema trunk (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (2)
Fatigue (General disorders) | 80 (279)
Fever (General disorders) | 19 (29)
Flu like symptoms (General disorders) | 3 (4)
Gen disord and admin site conds-Oth spec (General disorders) | 7 (11)
Injection site reaction (General disorders) | 6 (8)
Localized edema (General disorders) | 1 (1)
Malaise (General disorders) | 4 (7)
Non-cardiac chest pain (General disorders) | 18 (27)
Pain (General disorders) | 13 (20)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 9 (9)
Lung infection (Infections and infestations) | 3 (3)
Mucosal infection (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 5 (5)
Otitis media (Infections and infestations) | 2 (2)
Papulopustular rash (Infections and infestations) | 1 (3)
Paronychia (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 6 (7)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 11 (17)
Urinary tract infection (Infections and infestations) | 2 (4)
Vaginal infection (Infections and infestations) | 2 (4)
Bruising (Injury, poisoning and procedural complications) | 3 (7)
Dermatitis radiation (Injury, poisoning and procedural complications) | 5 (5)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (7)
Alanine aminotransferase increased (Investigations) | 34 (66)
Alkaline phosphatase increased (Investigations) | 12 (13)
Aspartate aminotransferase increased (Investigations) | 23 (35)
Blood bilirubin increased (Investigations) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 3 (8)
CO diffusing capacity decreased (Investigations) | 4 (9)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Forced expiratory volume decreased (Investigations) | 1 (1)
Hemoglobin increased (Investigations) | 2 (3)
INR increased (Investigations) | 2 (4)
Investigations - Other, specify (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 54 (228)
Lymphocyte count increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 94 (468)
Platelet count decreased (Investigations) | 21 (56)
Vital capacity abnormal (Investigations) | 2 (3)
Weight gain (Investigations) | 8 (20)
Weight loss (Investigations) | 4 (12)
White blood cell decreased (Investigations) | 93 (459)
Anorexia (Metabolism and nutrition disorders) | 25 (47)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 28 (63)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 (35)
Hypocalcemia (Metabolism and nutrition disorders) | 15 (25)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 17 (33)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 9 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (35)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (32)
Bone pain (Musculoskeletal and connective tissue disorders) | 10 (12)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (5)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (5)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 3 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (39)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (30)
Akathisia (Nervous system disorders) | 2 (4)
Amnesia (Nervous system disorders) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 2 (6)
Concentration impairment (Nervous system disorders) | 1 (4)
Dizziness (Nervous system disorders) | 15 (25)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 11 (31)
Headache (Nervous system disorders) | 30 (62)
Memory impairment (Nervous system disorders) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 3 (4)
Neuralgia (Nervous system disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 6 (12)
Peripheral motor neuropathy (Nervous system disorders) | 9 (23)
Peripheral sensory neuropathy (Nervous system disorders) | 42 (103)
Seizure (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 19 (55)
Depression (Psychiatric disorders) | 5 (9)
Insomnia (Psychiatric disorders) | 22 (64)
Irritability (Psychiatric disorders) | 1 (5)
Libido decreased (Psychiatric disorders) | 2 (5)
Restlessness (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (2)
Renal hemorrhage (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 6 (12)
Urinary tract pain (Renal and urinary disorders) | 2 (4)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 2 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 60 (125)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 50 (115)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 18 (23)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12 (16)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 38 (109)
Body odor (Skin and subcutaneous tissue disorders) | 1 (2)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (9)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 3 (10)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (7)
Nail ridging (Skin and subcutaneous tissue disorders) | 2 (4)
Photosensitivity (Skin and subcutaneous tissue disorders) | 4 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (29)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (14)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (23)
Scalp pain (Skin and subcutaneous tissue disorders) | 2 (7)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 12 (19)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 9 (19)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2)
Flushing (Vascular disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 7 (14)
Hypertension (Vascular disorders) | 11 (37)
Hypotension (Vascular disorders) | 4 (5)
Phlebitis (Vascular disorders) | 6 (13)
Superficial thrombophlebitis (Vascular disorders) | 5 (10)
Thromboembolic event (Vascular disorders) | 5 (11)
Vascular disorders - Other, specify (Vascular disorders) | 2 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT01118026/Prot_SAP_000.pdf